CLINICAL TRIAL: NCT04171960
Title: Clinical Evaluation of the i-STAT TBI Test
Status: Completed | Type: Observational
Sponsor: Abbott Point of Care (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CS-2018-0009
Record Dates: First submitted 2019-10-31; First posted 2019-11-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury
Keywords: i-STAT; Traumatic Brain Injury; Biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection; Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens retained for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Acute Blood Biomarker Branch: Blood drawn within 12 hours or 12-24 hours following injury for i-STAT TBI Testing and in-person baseline outcome assessments.
  Interventions: Diagnostic Test: Blood draw; Other: Outcome assessments

INTERVENTIONS:
Diagnostic Test: Blood draw — Venous whole blood collection within 12 hours and 12-24 hours following injury.
Other: Outcome assessments — Administered at baseline.

SUMMARY:
The goal of this study is to evaluate the i-STAT TBI test to assist determining the need for a computed tomography (CT) scan in patients with suspected mild traumatic brain injury (TBI).

Patients will be asked to provide a blood sample.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical performance of the i-STAT TBI test for the proposed intended use; to assist in determining the need for a computed tomography (CT) scan in patients presenting with suspected mild traumatic brain injury (TBI) who are 18 years of age or older.

The secondary objective of this study is the collection of additional data and specimens from all study subjects that may support other purposes related to the understanding of TBI.

ELIGIBILITY:
Acute Blood Biomarker Branch Subject Inclusion Criteria:

1. 18 years of age or older.
2. Subject or Legally Authorized Representative (LAR) provided informed consent for the Acute Blood Biomarker Branch (waiver of consent may be acceptable, per IRB).
3. Subject presented to a health care facility or emergency department with a suspected TBI resulting from an insult to the head by an external force within 12 hours of the injury.
4. Subject has a CT scan of the head with all sequences (bone and soft tissue) ordered as part of standard of care at the enrolling facility or are transferred to the enrolling facility with a head CT scan sent from the originating facility.
5. As a result of this head injury, the subject has sustained a traumatically induced physiological disruption of brain function, as manifested by at least one of the following.

   1. Any period of loss of consciousness
   2. Any loss of memory for events immediately before or after the injury
   3. Any alteration of mental state at the time of the injury
   4. Focal neurological deficits that may or may not be transient

Acute Blood Biomarker Branch Subject Exclusion Criteria.

1. Previous enrollment in this study
2. Current (on-going) enrollment in a therapeutic or interventional clinical trial (drug or device)
3. Primary diagnosis at the enrolling facility of ischemic or hemorrhagic stroke
4. Time of injury is unknown and cannot be estimated
5. Presented with penetrating head trauma or spinal cord injury (American Spinal Injury Association [ASIA] score of C or worse) at the enrolling facility
6. Standard of care head CT scan procedures not completed prior to Emergency Department (ED) discharge
7. Prisoners or patients in custody
8. Patients on psychiatric hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of patients who are 18 years of age or older presenting to the Healthcare Facility with suspected mild TBI*, a GCS score of 13-15 and within 24 hours of head injury.
  *TBI includes the head being struck or striking an object, or the brain undergoing an acceleration/deceleration movement without direct external trauma to the head.
Sampling Method: Non-Probability Sample
Enrollment: 1106 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
i-STAT TBI Test relative to standard of care Computed Tomography (CT) findings. | Within 24 Hours of Traumatic Brain Injury (TBI)
  Results of the i-STAT TBI Test (elevated/not elevated) relative to CT findings (+/-) for intra-cranial lesions for each subject.
Clinical performance measurement of the i-STAT TBI Test. | Within 24 hours of Traumatic Brain Injury (TBI)
  Clinical performance metrics included, clinical sensitivity, clinical specificity, negative predictive value (NPV), positive predictive value (PPV), adjusted negative predictive value (adj. NPV) calculated to a 6% CT positive prevalence rate, negative likelihood ratio (neg. LR) and positive likelihood ratio (pos. LR).

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, MS, MBA, Study Director — Abbott Point of Care
Locations (21):
- United States (21):
  - University of California, San Francisco, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Craig Hospital, Englewood, Colorado
  - University of Miami, Miami, Florida
  - Rehabilitation Hospital of Indiana, Carmel, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Texas, Austin, Austin, Texas
  - University of Texas, South Western, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Sciences Center of Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Plan is currently undecided.

REFERENCES:
- [Background] Papa L, Brophy GM, Welch RD, Lewis LM, Braga CF, Tan CN, Ameli NJ, Lopez MA, Haeussler CA, Mendez Giordano DI, Silvestri S, Giordano P, Weber KD, Hill-Pryor C, Hack DC. Time Course and Diagnostic Accuracy of Glial and Neuronal Blood Biomarkers GFAP and UCH-L1 in a Large Cohort of Trauma Patients With and Without Mild Traumatic Brain Injury. JAMA Neurol. 2016 May 1;73(5):551-60. doi: 10.1001/jamaneurol.2016.0039. PMID 27018834
- [Background] Bazarian JJ, Biberthaler P, Welch RD, Lewis LM, Barzo P, Bogner-Flatz V, Gunnar Brolinson P, Buki A, Chen JY, Christenson RH, Hack D, Huff JS, Johar S, Jordan JD, Leidel BA, Lindner T, Ludington E, Okonkwo DO, Ornato J, Peacock WF, Schmidt K, Tyndall JA, Vossough A, Jagoda AS. Serum GFAP and UCH-L1 for prediction of absence of intracranial injuries on head CT (ALERT-TBI): a multicentre observational study. Lancet Neurol. 2018 Sep;17(9):782-789. doi: 10.1016/S1474-4422(18)30231-X. Epub 2018 Jul 24. PMID 30054151